CLINICAL TRIAL: NCT06996379
Title: Use of the J-Tip Needle-Free Injection System With 1% Lidocaine to Reduce Paracentesis-Related Discomfort
Brief Title: J-Tip Use for Paracentesis in Adults With Liver Cirrhosis and Ascites
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Emily Kahn, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00222556
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Evaluate Patient Comfort Level During Paracentesis by Numbing Skin With a Needle-less Device, Instead of Using a Needle to Numb the Skin
Keywords: J-Tip; needle-less device; needle-free device; paracentesis; comfort; numbing; level of comfort; procedure-related pain

STUDY DESIGN:
Intervention Model Description: Upon enrollment, patients will be randomized using a randomization module built into the REDCap project, to either the control (25-gauge needle) or J-Tip arm. Patients will undergo diagnostic and/or therapeutic ultrasound-guided paracentesis as per standard of practice. The only difference between the groups will be the method of administering the superficial (intradermal) anesthesia. Based on randomization, lidocaine will be administered superficially via either 25 gauge intradermal needle (control) or the J-tip Needle-Free injection system. Following this superficial anesthesia injection, both groups will receive deeper subcutaneous lidocaine via a second 22-gauge needle per standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (25-gauge Needle) Arm, Current Standard of Care (Other): During abdominal paracentesis lidocaine will be administered superficially (intradermally) via a 25-gauge intradermal needle (control), as per the current standard of care.
  Interventions: Device: Control (Standard treatment)
- Experimental (J-Tip device) Arm (Experimental): During abdominal paracentesis lidocaine will be administered superficially (intradermally) via needle-free injection system (the J-Tip device). This is the experimental arm to compare to the 25-gauge needle (standard of care) method of intradermal lidocaine administration during abdominal paracentesis.
  Interventions: Device: Experimental J-Tip Needle-Free Injection System

INTERVENTIONS:
Device: Experimental J-Tip Needle-Free Injection System — This experimental intervention arm will include use of the J-Tip needle-less device to administer a one-time dose of 1% lidocaine during the superficial (intradermal) numbing step of a bedside abdominal paracentesis for adults with cirrhosis of the liver and ascites requiring bedside paracentesis.
  Other Names: J-Tip; J-Tip device; J-Tip needle-less device; J-Tip needle-free device
  Arms: Experimental (J-Tip device) Arm
Device: Control (Standard treatment) — The control intervention arm will include use of a 25-gauge needle (standard of care) to administer a one-time dose of 1% lidocaine during the superficial (intradermal) numbing step of a bedside abdominal paracentesis for adults with cirrhosis of the liver and ascites requiring bedside paracentesis.
  Other Names: control; 25-gauge needle
  Arms: Control (25-gauge Needle) Arm, Current Standard of Care

SUMMARY:
The purpose of this clinical trial is to evaluate the level of comfort adult patients with cirrhosis of the liver and ascites presenting to Northwestern Memorial Hospital experience during a bedside abdominal paracentesis by numbing the skin with a needle-less device (the J-Tip), instead of using a needle to numb the skin. The main questions it aims to answer are the J-Tip effect upon:

1. Pain during intra-dermal local anesthetic administration
2. Pain during subcutaneous local anesthetic administration
3. Pain during paracentesis
4. Procedure-related anxiety

Participants will be randomly assigned to have their skin numbed either in the usual way with a needle or with the J-Tip. Participants will be responsible for having a paracentesis done in their hospital room and answering the survey questions regarding pain experienced during the procedure and how they would feel if they needed to have this procedure performed again. There is also a telephone follow-up survey 2 days after the procedure to ask the participant about their experience post-procedure. We will also collect data about any procedure complications.

DETAILED DESCRIPTION:
The investigators would like to conduct an open label randomized control trial quantifying perception of pain during both administration of local anesthetic and during abdominal paracentesis when superficial (intradermal) lidocaine is administered via needle-free injection system as compared to via 25-gauge needle (standard of care). The study will include at least 110 participants in the emergency room or admitted to a general medical service with cirrhosis and ascites requiring bedside paracentesis, including both diagnostic (only a small sample of fluid removed for testing) and/or therapeutic paracentesis (a large amount of fluid removed to relieve discomfort). The primary physician caring for the patient will determine whether a paracentesis is required (not the study investigators).

Patients ≥ 18 years of age presenting to Northwestern Memorial Hospital with cirrhosis of the liver and ascites who require bedside paracentesis will be eligible for this study. Eligible patients will be identified by Emergency Department and Hospital Medicine providers who will notify study investigators. Upon identifying the patients and confirming eligibility through reviewing patients' charts and verbal screening questions, a study team member will approach patients, explain the study, and obtain written informed consent for those patients willing to participate. Patients whose preferred language is not English, those who have previously received or are currently receiving chemotherapy (as the J-Tip is contra-indicated in patients receiving chemotherapy), and those who are otherwise unable to provide informed consent will be excluded. Pregnant patients, prisoners, or other detained individuals will be excluded as well.

Upon enrollment, patients will be randomized using a randomization module built into the REDCap project, to either the control (25-gauge needle) or J-Tip arm. Patients will undergo diagnostic and/or therapeutic ultrasound-guided paracentesis as per standard of practice. The only difference between the groups will be the method of administering the superficial (intradermal) anesthesia. Based on randomization, lidocaine will be administered superficially via either 25-gauge intradermal needle (control) or the J-tip Needle-Free injection system. Following this superficial anesthesia injection, both groups will receive deeper subcutaneous lidocaine via a second 22-gauge needle per standard of care.

Following the procedure, the patient will be asked by a study coordinator (in person or over the phone) to rate their pain using a numeric rating scale (NRS from 1 to 10; 0= no pain, 10 = extreme pain). Patients will also be asked about anticipated anxiety during future procedures. The thickness of skin tissue and tissue deep to the skin (subcutaneous tissue) overlying the ascites fluid in millimeters as measured by ultrasound will also be measured by the study investigators (Dr. Kahn or Dr. Barsuk) and recorded. Drs. Kahn and Barsuk are on the Hospital Medicine Procedure Service and are routinely consulted to perform paracentesis procedures on patients.

Two days following the procedure, a study member will contact the patient (in person or via phone) to inquire about complications including bleeding/bruising and pain following the procedure. Dr. Kahn will also chart review to assess for hemodynamically significant bleed or procedure related complication.

ELIGIBILITY:
Inclusion Criteria:

- Adult (age > 18 years) patients in the emergency department or admitted to the general medical service at Northwestern Memorial Hospital who:

1. Have cirrhosis and ascites
2. Require diagnostic and/or therapeutic paracentesis as determined by their primary physician
3. Have capacity as determined by their ED or inpatient provider to consent for the procedure

c. Speak English as a preferred language

Exclusion Criteria:

* Have ever received chemotherapy, as this is a contra-indication to J-Tip use
* Lack capacity to consent for the procedure and/or capacity to rate their pain using the numeric pain rating scale
* Have a contraindication to bedside paracentesis, including:

  1. Procedure deemed unsafe due to insufficient ascites/suboptimal location of ascites as evaluated by ultrasound
  2. Cellulitis overlying the site of aspiration
  3. Pregnancy
* Do not speak English as a preferred language
* Are prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Pain during intra-dermal (superficial) local anesthetic administration | From enrollment to end of procedure (approximately 2 hours).
  We seek to investigate the use of the J-Tip Needle-Free Injection System during bedside abdominal paracentesis in improving patient tolerance of the local anesthetic process and the procedure. Following the procedure, the patient will be asked by a study coordinator (in person or over the phone) to rate their pain using a numeric rating scale (NRS from 1 to 10; 0= no pain, 10 = extreme pain).
Pain during subcutaneous local anesthetic administration | From enrollment to end of procedure (approximately 2 hours).
  We seek to investigate the use of the J-Tip Needle-Free Injection System during bedside abdominal paracentesis in improving patient tolerance of the local anesthetic process and the procedure. Following the procedure, the patient will be asked by a study coordinator (in person or over the phone) to rate their pain using a numeric rating scale (NRS from 1 to 10; 0= no pain, 10 = extreme pain).
Pain during paracentesis | From enrollment to end of procedure (approximately 2 hours).
  We seek to investigate the use of the J-Tip Needle-Free Injection System during bedside abdominal paracentesis in improving patient tolerance of the local anesthetic process and the procedure. Following the procedure, the patient will be asked by a study coordinator (in person or over the phone) to rate their pain using a numeric rating scale (NRS from 1 to 10; 0= no pain, 10 = extreme pain).

SECONDARY OUTCOMES:
Anxiety about future procedures | From enrollment to end of procedure (approximately 2 hours).
  We seek to investigate the use of the J-Tip Needle-Free Injection System during bedside abdominal paracentesis in improving patient tolerance of the local anesthetic process and the procedure. Patients will be asked about anticipated anxiety during future procedures.
Procedure related complications | From enrollment to end of telephone follow-up survey (approximately 2 days).
  We seek to investigate the use of the J-Tip Needle-Free Injection System during bedside abdominal paracentesis in improving patient tolerance of the local anesthetic process and the procedure. Two days following the procedure, a study member will contact the patient (in person or via phone) to inquire about complications including bleeding/bruising and pain following the procedure. Dr. Kahn will also chart review to assess for hemodynamically significant bleed or procedure related complication.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Kahn, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hajimaghsoudi M, Vahidi E, Momeni M, Arabinejhad A, Saeedi M. Comparison of local anesthetic effect of lidocaine by jet injection vs needle infiltration in lumbar puncture. Am J Emerg Med. 2016 Jul;34(7):1225-9. doi: 10.1016/j.ajem.2016.03.030. Epub 2016 Mar 16. PMID 27055606
- [Background] Gozdemir M, Demircioglu RI, Karabayirli S, Sert H, Muslu B, Usta B, Yazici U. A Needle-Free Injection System (INJEX) with lidocaine for epidural needle insertion: A randomized controlled trial. Pak J Med Sci. 2016 May-Jun;32(3):756-61. doi: 10.12669/pjms.323.9174. PMID 27375728
- [Background] Gursoy A, Ertugrul DT, Sahin M, Tutuncu NB, Demirer AN, Demirag NG. Needle-free delivery of lidocaine for reducing the pain associated with the fine-needle aspiration biopsy of thyroid nodules: time-saving and efficacious procedure. Thyroid. 2007 Apr;17(4):317-21. doi: 10.1089/thy.2006.0326. PMID 17465861
- [Background] Burns CA, Ferris G, Feng C, Cooper JZ, Brown MD. Decreasing the pain of local anesthesia: a prospective, double-blind comparison of buffered, premixed 1% lidocaine with epinephrine versus 1% lidocaine freshly mixed with epinephrine. J Am Acad Dermatol. 2006 Jan;54(1):128-31. doi: 10.1016/j.jaad.2005.06.043. PMID 16384767
- [Background] Duncanson E, Le Leu RK, Shanahan L, Macauley L, Bennett PN, Weichula R, McDonald S, Burke ALJ, Collins KL, Chur-Hansen A, Jesudason S. The prevalence and evidence-based management of needle fear in adults with chronic disease: A scoping review. PLoS One. 2021 Jun 10;16(6):e0253048. doi: 10.1371/journal.pone.0253048. eCollection 2021. PMID 34111207